CLINICAL TRIAL: NCT03536221
Title: D2D What is the Prevalence of Female Pelvic Floor Disorders in Minnesota?
Brief Title: What is the Prevalence of Female Pelvic Floor Disorders in Minnesota?
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00003436
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Prolapse; Urinary Incontinence; Fecal Incontinence; Bladder Pain Syndrome
MeSH Terms: conditions — Prolapse; Urinary Incontinence; Fecal Incontinence; Cystitis, Interstitial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine the prevalence of pelvic organ prolapse and urinary incontinence among women in Minnesota using a short web-based self-administered questionnaire.

DETAILED DESCRIPTION:
The study will be administered at the 2018 Minnesota State Fair at the Driven to Discover building. The study will be administered entirely for research purposes. All data will be self-reported (see attached survey). Data collection will be through a web-based version of the EPIQ loaded into Research Electronic Data Capture REDCap, a secure web-based system for data collection. Data collection will occur over 6 half day sessions at the University of Minnesota D2D building at the Minnesota State Fair Grounds while the Fair is running.

ELIGIBILITY:
Inclusion Criteria:

* Women who are age 18 or older on the date they take the survey who are willing to take the survey. Pregnant women may participate in the survey.

Exclusion Criteria:

* Inability to provide consent to take the survey, and inability to speak and understand English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women aged 18 years and older who attend the Minnesota State Fair and are willing to participate in the survey.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Prolapse | Aug-Sep 2018
  Prevalence of prolapse in the population studied
Urinary incontinence | Aug-Sep 2018
  Prevalence of urinary incontinence in the population studied
Fecal incontinence | Aug-Sep 2018
  Prevalence of fecal incontinence in the population studied
Bladder pain | Aug-Sep 2018
  Prevalence of bladder pain in the population studied

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided
No plan at present

REFERENCES:
- [Background] Egger MJ, Lukacz ES, Newhouse M, Wang J, Nygaard I. Web versus paper-based completion of the epidemiology of prolapse and incontinence questionnaire. Female Pelvic Med Reconstr Surg. 2013 Jan-Feb;19(1):17-22. doi: 10.1097/SPV.0b013e31827bfd93. PMID 23321654
- [Result] Olsen AL, Smith VJ, Bergstrom JO, Colling JC, Clark AL. Epidemiology of surgically managed pelvic organ prolapse and urinary incontinence. Obstet Gynecol. 1997 Apr;89(4):501-6. doi: 10.1016/S0029-7844(97)00058-6. PMID 9083302
- [Result] Wu JM, Kawasaki A, Hundley AF, Dieter AA, Myers ER, Sung VW. Predicting the number of women who will undergo incontinence and prolapse surgery, 2010 to 2050. Am J Obstet Gynecol. 2011 Sep;205(3):230.e1-5. doi: 10.1016/j.ajog.2011.03.046. Epub 2011 Apr 2. PMID 21600549
- [Result] Lukacz ES, Lawrence JM, Buckwalter JG, Burchette RJ, Nager CW, Luber KM. Epidemiology of prolapse and incontinence questionnaire: validation of a new epidemiologic survey. Int Urogynecol J Pelvic Floor Dysfunct. 2005 Jul-Aug;16(4):272-84. doi: 10.1007/s00192-005-1314-5. Epub 2005 Apr 26. PMID 15856132
- See also: Predicted growth of Minnesota's population — https://mn.gov/admin/demography/data-by-topic/population-data/our-estimates/
- See also: Age breakdown of Minnesota's predicted growth — https://mn.gov/admin/demography/data-by-topic/aging/